CLINICAL TRIAL: NCT00173953
Title: Lymphocytic Subsets and Cytokine Production in the Gastric Samples of Patients With Helicobacter Pylori Infection
Brief Title: Lymphocytic Subsets and Cytokine Production With H. Pylori Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 90M010; 90M010
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2000-12

CONDITIONS: Duodenal Ulcer; Gastric Ulcer; Dyspepsia
Keywords: H. pylori、immune response、lymphocytic subsets、cytokine
MeSH Terms: conditions — Duodenal Ulcer; Stomach Ulcer; Dyspepsia | interventions — Immunity

INTERVENTIONS:
Procedure: immune response

SUMMARY:
The aims of this study are 1) to determine the cytokines produced by both Th1 and Th2 subsets in gastric antral biopsy specimens from Taiwanese patients before and after anti H. pylori therapy; 2) to obtain a detailed phenotypic characterization and distribution pattern of mucosal lymphocytes in H. pylori-associated gastritis and to define possible contributing immune mechanisms responsible for the chronicity of the disease and its associated lesions.

DETAILED DESCRIPTION:
Helicobacter pylori, a Gram-negative spiral bacterium, has been first isolated from a patient with chronic active gastritis since 1982. Recent studies strongly suggest that chronic infection with H. pylori is tightly associated with chronic gastritis, peptic ulcer, and gastric carcinoma. However, only a minority of infected people develop signs and symptoms of gastric pathology. Thus, both host and microbial factors may lead to different outcomes of infection. In spite of high prevalence in general population and increasing clinical attention has been paid on this infection, the knowledge of pathogenic mechanism of H. pylori infection is still limited and little is known about the role of host immune response in the pathogenesis of disease.The aims of this study are 1) to determine the cytokines produced by both Th1 and Th2 subsets in gastric antral biopsy specimens from Taiwanese patients before and after anti H. pylori therapy; 2) to obtain a detailed phenotypic characterization and distribution pattern of mucosal lymphocytes in H. pylori-associated gastritis and to define possible contributing immune mechanisms responsible for the chronicity of the disease and its associated lesions.

ELIGIBILITY:
Inclusion Criteria:

* H. pylori infection

Exclusion Criteria:

* none

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2001-01; Study Completion 2001-10

PRIMARY OUTCOMES:
Cytokines produced by both Th1 / Th2 subsets in gastric antral biopsy specimens from Taiwanese patients before and after anti H. pylori therapy.

SECONDARY OUTCOMES:
Obtain a detailed phenotypic characterization and distribution pattern of mucosal lymphocytes in H. pylori-associated gastritis and to define immune mechanisms responsible for the chronicity of the disease and its associated lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Chin Yang, M.D., Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- Department of Internal Medicine, National Taiwan University Hospital, Taipei, Taiwan